CLINICAL TRIAL: NCT01346280
Title: Quality of Care: The Impact of Multidisciplinary Care on Processes and Outcomes of Cancer Care
Brief Title: Evaluation of Cancer Care Coordination in the National Cancer Institutes Community Cancer Center Programs
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911145; 11-C-N145
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-10-05

CONDITIONS: Non-Small Cell Lung Cancer (Stage III); Colon Cancer (Stage II &Amp; III); Rectal Cancer (Stage III)
Keywords: Adherence to Evidence-Based Guidelines; Multidisciplinary Care; Patient Experiences; Quality of Care Outcomes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

-Coordinated cancer care provided by doctors, nurses, social workers, and other care providers is believed to improve patient and physician satisfaction and patient evaluation for enrollment in clinical trials. But no research has been done to show that this approach improves patient experiences and outcomes. Researchers want to study this model to better understand how it can improve cancer treatment and patient outcomes.

Objectives:

- To assess the relationship between coordinated care and cancer treatment processes and outcomes.

Eligibility:

- Individuals who are at least 18 years of age. Those who take part must have been diagnosed with colon, rectal, or non-small-cell lung cancer. They also must be receiving or have been treated at one of the 16 NCI Community Cancer Center program sites.

Design:

* Researchers will collect medical records data from participants.
* Participants will complete a questionnaire about 8 weeks after the end of all planned cancer treatment. They will be asked questions about their experience with coordinated cancer care. They will also be asked for any comments or concerns they had during and after treatment.
* No treatment or additional tests will be provided as part of this protocol.

DETAILED DESCRIPTION:
There is little evidence regarding the effect of multidisciplinary care (MDC) on health outcomes across various cancer sites, including colon, rectal, and lung cancer. The current study addresses this gap by providing preliminary data regarding the relationship between MDC and selected processes and outcomes of care in NCCCP pilot sites. The long-term goal of this preliminary study is to generate effect sizes, establish feasibility, and build infrastructure to support the development of a larger more definitive study of MDC outcomes. The key aim of this pilot study is to determine the relationship between specific MDC assessment areas identified by a pre-existing MDC assessment tool (http://ncccp .cancer.gov /NCCCPMDC- Matrix- Tool. pdf ): case planning, physician engagement, coordination of care, infrastructure, financial, clinical trials and medical records, and each of the following outcomes [0] and processes [P]: 1) time to receipt of initial therapy[P]; 2) receipt of multi-modality therapy[O]; 3) evaluation for enrollment in a clinical trial[P]; 4) patient experience[O]; 5) adherence to NCCN treatment guidelines[P]; and 6) all-cause survival[O]. The study focuses on adult patients with an incident diagnosis of Stage III colon cancer, Stage II or III rectal cancer, or Stage III non-small cell lung cancer.

We will quantify the relationship between MDC, various care processes and outcomes across 16 participating NCCCP sites, testing the hypothesis that increasing levels of MDC identified by the MDC tool are associated with improvement in care quality and a survival advantage.

Significant progress has been achieved in the past year establishing the necessary

processes for conducting the research study and the deliverables associated with the study. In terms of process outcomes, we can report the following:

1. Institutional Review Board approval for the multidisciplinary care study at all 16

   sites;
2. The development of a Standard Operating Procedures manual for use by the 16 sites;
3. The development of a data collection form (Site Data Collection Tool) to be used for

   collecting information that is not available via the pre-existing web-based data

   collection system that is in place at the 16 sites;
4. The development of a data collection form to be used for documenting the facility s

   annual scores using the Multidisciplinary Care Assessment tool.
5. The development of a flowchart for use in operationalizing the measurement of

   NCCN guideline adherence for patients with Stage III non small cell lung cancer;
6. The development of a Frequently Asked Questions document to assist with

   addressing questions in real time;
7. Multiple training sessions/webinars have been held for the participating sites.
8. Monthly conference call with the research team and representatives from all

participating sites.

ELIGIBILITY:
* INCLUSION CRITERIA:

Stage III colon cancer, Stage II or III rectal cancer or Stage III lung cancer. Additional inclusion criteria: Age: equal to or greater than 18 at time of diagnosis; English speaking (native or non-native); First or only cancer diagnosis; All or part of first course of treatment was performed at the reporting facility.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1079 (Actual)
Dates: Start 2011-04-16; Study Completion 2015-10-05

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Castro, R.N., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Freeman RK, Van Woerkom JM, Vyverberg A, Ascioti AJ. The effect of a multidisciplinary thoracic malignancy conference on the treatment of patients with lung cancer. Eur J Cardiothorac Surg. 2010 Jul;38(1):1-5. doi: 10.1016/j.ejcts.2010.01.051. Epub 2010 Mar 4. PMID 20206544
- [Background] Fennell ML, Das IP, Clauser S, Petrelli N, Salner A. The organization of multidisciplinary care teams: modeling internal and external influences on cancer care quality. J Natl Cancer Inst Monogr. 2010;2010(40):72-80. doi: 10.1093/jncimonographs/lgq010. PMID 20386055
- [Background] Sidhom MA, Poulsen MG. Multidisciplinary care in oncology: medicolegal implications of group decisions. Lancet Oncol. 2006 Nov;7(11):951-4. doi: 10.1016/S1470-2045(06)70942-1. PMID 17081921